CLINICAL TRIAL: NCT02230007
Title: Contribution of the MEOPA in the Physiotherapy Care of Painful Articular Steepness Among Elderly
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2013-000065-37; 12AOI02 (Other: CHU DE NICE)
Record Dates: First submitted 2013-05-07; First posted 2014-09-03 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2013-12

CONDITIONS: Pain Management and Care
MeSH Terms: conditions — Agnosia | interventions — Meopa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MEOPA (Experimental): ENTONOX (MEOPA)gas Duration of treatment of a subject according to the protocol: 60 MINUTES Inhalation use
  Interventions: Drug: MEOPA
- Without MEOPA (No Intervention): Physiotherapit care without MEOPA

INTERVENTIONS:
Drug: MEOPA — 3 sessions of reeducation using MEOPA
  Arms: MEOPA

SUMMARY:
The MEOPA is used to obtain an analgesia of the short-term painful acts. To the population of elderly patients, the therapeutic resources to control the passing pain require in their manipulation a certain caution and are not divested of side effects badly tolerated at this age. An alternative in the opioid presents all its interest. The MEOPA is here an alternative of choice in the care of these pains, in particular in case of pre-existent cognitive achievement, of polypathologies or of polymédication.

The gas MEOPA administered to the mask could thus be an effective additive in the physiotherapy treatment of the elderly person.

The main objective is to Assess the efficacy , in terms of recovery of the hip and knee joint articular amplitude, of 3 sessions of reeducation using MEOPA versus standard reeducation within a population of elderly patients presenting a pain during the physiotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 65 years old or more
* Patients having a prescription for physiotherapy
* Absence of contraindication to MEOPA
* Patients whose initial assessment show a passive articular deficit of at least a joint of hip or the knee and whose painful assessment is ≥ 5 or ≥ 2 during mobilisation on the validated scale Algoplus
* Patients whose reeducation project established by the physiotherapist
* Patients having agreed to participate in the study and having signed the consent
* Subjects affiliated to the social security system

Exclusion Criteria:

* Patient requiring a ventilation in pure oxygen
* Patient with a consciousness deterioration preventing his cooperation
* Care under MEOPA during the period of the protocol and during the month which precedes
* Increase of the dosage of morphine of less than 48 hours Patient under guardianship

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-05 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
% of recovery of the hip and knee joint articular amplitude | 5 days
  % of recovery of the hip and knee joint articular amplitude during 5 days after 3 sessions of reeducation using MEOPA versus standard reeducation within a population of elderly patients presenting a pain during the physiotherapy treatment; measure % of recovery of the hip and knee joint articular amplitude two times : before the beginning of the session of reeducation and at the end of the session

SECONDARY OUTCOMES:
Measure of the pain | 5 days
  Patient answer a questionnaire on his pain at the beginning of each session of reeducation (5 sessions)
Patients'satisfaction | End of the period of care (up to 5 days)
  Patient answer a questionnaire on this satisfaction at the end of the period of care of the protocol.
Physiotherapists'satisfaction | End of all the period of care (up to 5 days)
  Physiotherapists answer a questionnaire on this satisfaction of the use of the MEOPA

CONTACTS AND LOCATIONS:
Overall Officials: Véronique Mailland, MD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (2):
- France (2):
  - Pôle de Gérontologie Hôpital de Cimiez CHU de Nice, Nice
  - CHU de Nice, Nice